CLINICAL TRIAL: NCT01037933
Title: Comedy in Chemotherapy (COMIC) Study
Acronym: COMIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Collaborators: Queen Emma Nursing Research Institute (Unknown); University of Hawaii (Other)
Responsible Party: Hob Osterlund, APRN Clinical Nurse Specialist, Pain and Palliative Care Department, The Queen's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RA2007020; Hob Osterlund
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Cancer; Chemotherapy
Keywords: Cancer; Humor; Distraction; Comedy; Chemotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Humor intervention (Active Comparator): A 45-minute humorous DVD ("Bananas Bunch") using a portable DVD player.
  Interventions: Other: Humor intervention
- Non-humor intervention (Active Comparator): A 45-minute non-humorous DVD "The A to Z of Steam Railways" using a portable DVD player.
  Interventions: Other: Non-humor intervention (distraction)

INTERVENTIONS:
Other: Humor intervention — A 45-minute humorous DVD ("Bananas Bunch") using a portable DVD player.
  Arms: Humor intervention
Other: Non-humor intervention (distraction) — A 45-minute non-humorous DVD ("The A to Z of Steam Railways") using a portable DVD player
  Arms: Non-humor intervention

SUMMARY:
Primary aims: To compare changes in (a) symptoms related to cancer and chemotherapy, (b) a marker of immune function (salivary immunoglobulin A), and (c) a hormonal marker of emotional stress (salivary cortisol) between two groups of patients who view a humorous or non-humorous DVD.

Secondary aim: To describe the perception of patients, caregivers, and nurses regarding the overall intervention experience.

DETAILED DESCRIPTION:
Patients were recruited from the Outpatient Oncology (OPO) clinic at QMC. After signing an informed consent, patients receiving intravenous chemotherapy were randomly assigned to view a 45-minute humorous DVD or non-humorous DVD. The following measurements were obtained before and after patients viewed the DVD: Edmonton Symptom Assessment Scale (ESAS) and the state portion of the Spielberger State-Trait Anxiety Index (STAI-S) to assess symptoms related to cancer and chemotherapy, salivary immunoglobulin A (IgA) to assess immune function and salivary cortisol to assess emotional stress. In addition, patients, caregivers, and nurses were asked open-ended questions after the intervention to ascertain their impression of the overall intervention experience. Multiple analysis of covariance (MANCOVA) were be used to analyze changes in ESAS, STAI-S, IgA and cortisol within and between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cancer
2. Receiving intravenous chemotherapy in the OPO clinic at QMC
3. Has a minimum appointment time in OPO of two hours
4. Age 21 or older
5. Speaks English

Exclusion Criteria:

1. Blind
2. Deaf
3. Diagnosis of head/neck cancer
4. Severe oral mucositis
5. Cognitively impaired

   -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To compare changes in symptoms related to cancer and chemotherapy after a humor vs. non-humor intervention | One day

SECONDARY OUTCOMES:
To compare changes in a marker of immune function (salivary immunoglobulin A), and a hormonal marker of emotional stress (salivary cortisol) between two groups of patients who view a humorous or non-humorous DVD. | One day

CONTACTS AND LOCATIONS:
Overall Officials: Hob Osterlund, RN, MS, Principal Investigator — The Queen's Medical Center; Brad Willcox, MD, Study Director — The Queen's Medical Center
Locations (1):
- The Queen's Medical Center, Honolulu, Hawaii, United States

REFERENCES:
- See also: The Queen's Medical Center — http://queens.org